CLINICAL TRIAL: NCT06538948
Title: Direct Measurement of Ingestive Behaviour in Relation to Sex Differences and Gastrointestinal Hormone Levels in Patients After Metabolic and Bariatric Surgery
Acronym: DIBASH
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Florida State University (Other); University College Dublin (Other)
Responsible Party: Principal Investigator, Marco Bueter, Head of Bariatric Surgery, University of Zurich
Other Study IDs: 2023-02109
Record Dates: First submitted 2024-07-25; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Obesity
Keywords: Obesity; Ingestive Behaviour; Bariatric Surgery; Gut Hormones; Drinkometer
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples are collected from venous blood before, directly after, 30, and 90 minutes after the meal test. Plasma samples will be isolated from blood samples and stored at -80° C for later analysis. The analysis of DNA is not planned in this study. Nevertheless, plasma can contain cell-free DNA (cfDNA). Considering that no solution for the stabilisation of nucleic acid is added to the plasma samples, a complete or meaningful sequencing of the cfDNA can hardly be expected from the plasma samples collected in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Adult Females planned for RYGB surgery: Adult females leaving with obesity with BMI between 35 and 50 kg/m2 and scheduled for Roux-en-Y Gastric Bypass Surgery
  Interventions: Procedure: Bariatric Surgery
- Adult Females planned for SG surgery: Adult females leaving with obesity with BMI between 35 and 50 kg/m2 and scheduled for Sleeve Gastrectomy Surgery
  Interventions: Procedure: Bariatric Surgery
- Adult Females with Obesity: Adult females leaving with obesity with BMI between 30 and 50 kg/m2 but not scheduled for any procedures of bariatric surgery
- Adult Females with Normal-Weight: Adult females with normal weight with BMI between 18.5 and 24.9 kg/m2
- Adult Males planned for RYGB surgery: Adult males leaving with obesity with BMI between 35 and 50 kg/m2 and scheduled for Roux-en-Y Gastric Bypass Surgery
  Interventions: Procedure: Bariatric Surgery
- Adult Males with Obesity: Adult males leaving with obesity with BMI between 30 and 50 kg/m2 but not scheduled for any procedures of bariatric surgery
- Adult Males with Normal-Weight: Adult males with normal weight with BMI between 18.5 and 24.9 kg/m2
- Adult Females and Males 5 years after RYGB surgery: Adult Females and Males who underwent RYGB surgery 5 years before study recruitment and study measurements
  Interventions: Procedure: Bariatric Surgery

INTERVENTIONS:
Procedure: Bariatric Surgery — The intervention is not assigned to the participant after recruitment in the study, rather the intervention is an inclusion criteria for participation in the study.
  Groups: Adult Females and Males 5 years after RYGB surgery; Adult Females planned for RYGB surgery; Adult Females planned for SG surgery; Adult Males planned for RYGB surgery

SUMMARY:
Bariatric surgery (BS), especially procedures like Sleeve Gastrectomy (SG) and Roux-en-Y gastric bypass (RYGB), is the most effective treatment for obesity. Yet, the exact mechanisms governing its effect are somewhat elusive, with current research mainly focusing on post-operative food intake outcomes based on self-reported data, which might not fully capture the nuanced changes in eating behaviours.

To address these gaps, our study plans to employ the newly developed "drinkometer", a device capable of analysing the intricate changes in drinking behaviour following BS. This tool promises to bring a more detailed perspective to the changes in ingestive behaviours, bypassing the inaccuracies of self-reporting methods. By expanding our research to encompass diverse patient demographics and examining potential links to physiological shifts like gut hormone level alterations, the study aims to provide a more rounded understanding of the long-term impacts of BS on eating behaviours.

DETAILED DESCRIPTION:
HYPOTHESIS AND PRIMARY OBJECTIVE

So far, studies of ingestive behaviour in humans have produced ambiguous results. Moreover, direct measurements of ingestive behaviour in humans after BS are still rare and the roles of sex and gut hormones, as well as their relevance for clinical outcome parameters, such as body weight loss, remain elusive. A comprehensive understanding of how a given intervention such as BS affects food intake requires a detailed analysis of the ingestive behaviour itself, not simply the measurement of the outcome of the behaviour. In other words, the information on how the food is consumed is equally or even more important than the information on how much food has been ingested.

This study employs the drinkometer methodology to perform direct measurements of ingestive behaviour in male and female human patients after SG and RYGB along with parallel measurements of postprandial gut hormone levels. Furthermore, this study investigates the clinical relevance of changes in ingestive behaviour by correlating microstructural parameters with body weight loss in a consecutive set of patients who received RYGB at the University Hospital Zurich five years before the time of recruitment.

Of note, the proposed experiments aim to test specific hypotheses regarding the behavioural mechanisms underlying potential changes in food intake after BS in humans. Thus, this research do not aim to identify how BS affects one or the other single microstructural parameters of eating or drinking. Instead, this study investigates how a given intervention that is known to substantially affect food intake behaviour - such as BS - alters the profile of a group of microstructural parameters of ingestive behaviour in humans. Given that ingestive behaviour represents the readout of the central nervous system mechanisms controlling energy intake (e.g., palatability, aversion, avoidance, satiation), the results of the proposed studies will inform the search for the underlying neural circuits in the brain that are specifically altered by BS. If there is no altered behaviour, there would be no point in investigating the underlying physiology. More specifically, this study aims to:

1. Investigate longitudinal changes and differences in the ingestive behaviour of female patients before and within one year after either primary RYGB or primary SG (Study 1).
2. Investigate a possible association between the ingestive behaviour and the prandial gut hormone levels of female patients before and within one year after either primary RYGB or SG (Study 1).
3. Investigate a possible difference between the ingestive behaviour of female and male patients before and within one year after primary RYGB (Study 2).
4. Investigate a possible association between the postoperatively achieved body weight loss of female and male patients 5 years after primary RYGB and ingestive behaviour (Study 3).
5. Investigate, in a subset of responders and non-responders to primary RYGB, a possible association between postprandial gut hormone levels of female and male patients 5 years after primary RYGB and ingestive behaviour (Study 3).

PRIMARY AND SECONDARY ENDPOINTS

In the research protocol, the primary and secondary outcomes specific to each of the three studies planned within the research project have been described. Recognising that each study has its unique objectives and hypotheses, the outcomes have been specified distinctly for each study to ensure clarity and focus in the research approach.

For each of the three studies, the primary outcomes are those key results that the study is primarily designed to assess. These are the main effects or findings that are anticipated to provide the most significant insights into the research questions. Secondary outcomes, while still important, are additional results that can be explored after answering the main research questions. These might provide supplementary information, support the primary outcomes, or offer insights into other areas related to the main research question.

By presenting these outcomes separately for each study, this study aims to provide a structured and transparent overview of the research intentions, allowing for a clear understanding of the objectives and measures in each specific part of the project. This approach not only aids in maintaining the focus and integrity of each study but also assists in the clear communication of the research goals and methods.

PROJECT DESIGN

The proposed studies will test key elements of ingestive behaviour and their relation to pre- and postprandial levels of gut hormones as well as sex differences after the two most frequently performed bariatric operations. They will thus provide useful information for planning and conducting future trials in the field, such as optimal recruitment and retention strategies, intervention delivery, data collection methods and adherence to study protocols. The proposed studies will further provide empirical estimates of effect sizes of bariatric surgery and long-term associations of ingestive behaviour with gut hormones for post-bariatric body weight loss. The potential outcomes of Studies 1, 2 and 3 are conceptually different. Nevertheless, the results of these studies will complement each other as well as our findings from previous studies, and can be used to calculate sample sizes for future trials.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year
* BMI ≥ 35 kg/m2 for patients with planned RYGB or SG operation
* BMI ≥ 30 kg/m2 for external controls affected by obesity but no planned RYGB or SG within the next 12 months, and
* BMI ≥ 18.5 kg/m2 and ≤ 24.9 kg/m2 for controls without obesity.

Exclusion Criteria:

* history of previous bariatric operations and/ or revisional surgery (e.g., alteration of limb lengths after primary RYGB),
* smoking,
* established diagnosis of type 1 or 2 diabetes mellitus, and
* polycystic ovary syndrome (PCOS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with obesity and scheduled for bariatric surgery are recruited consecutively at the outpatient clinic of bariatric surgery at the University Hospital Zurich.
  Participants with obesity not scheduled for surgery are recruited at the private clinic "Adimed" in Winterthur.
  Participants without obesity are recruited from students, employees and faculty of the Faculty of Medicine of the University of Zurich.
Sampling Method: Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Drinkometer Measurement of Microstructural Parameters of Ingestive Behaviour, such as Suck Energy Intake and Burst Energy Intake. | One year after bariatric surgery
  Difference of the eleven microstructural parameters of ingestive behaviour within the cohorts with intervention at the end of follow-up compared to baseline measurements and differences between the cohorts with intervention and the cohorts without intervention will be measured with a drinkometer device. The microstructural parameters of ingestive behaviour are: mean suck energy intake (kcal), mean suck duration (s), mean suck rate (kcal/s), mean suck maximal rate (kcal/s), burst number (n), burst energy intake (kcal), burst duration (s), burst rate (kcal/s), number of sucks per burst (n), inter-burst intervals (s), and inter-suck intervals (s). On this platform, a separate entry for the eleven microstructural parameters is not done to avoid redundancy in the description.
Effect of the Gut Hormones in Plasma on the Microstructural Parameters of Ingestive Behaviour Measured with the Drinkometer Device | One year after bariatric surgery
  This study investigates the effect of pre- and post-prandial levels of gut hormones on the eleven microstructural parameters of ingestive behavior. These are: mean suck energy intake (kcal), mean suck duration (s), mean suck rate (kcal/s), mean suck maximal rate (kcal/s), burst number (n), burst energy intake (kcal), burst duration (s), burst rate (kcal/s), number of sucks per burst (n), inter-burst intervals (s), and inter-suck intervals (s). On this platform, a separate entry for the eleven microstructural parameters is not done to avoid redundancy in the description. The study focuses on the influence of the following gut hormones: leptin, ghrelin, cholecystokinin (CCK), glucagon-like peptide-1 (GLP-1), gastric inhibitory polypeptide (GIP), amylin, peptide YY (PYY), and insulin. These hormone concentrations are measured both pre- and post-prandially in the blood and are expressed in their respective units of measure (e.g., leptin in ng/mL, ghrelin in pg/mL).
Effect of Biological Sex (Male or Female) on the Microstructural Parameters of Ingestive Behaviour Measured with the Drinkometer Device | One year after bariatric surgery
  This study investigates the effect of biological sex (male or female) on the eleven microstructural parameters of ingestive behavior. These parameters are: mean suck energy intake (kcal), mean suck duration (s), mean suck rate (kcal/s), mean suck maximal rate (kcal/s), burst number (n), burst energy intake (kcal), burst duration (s), burst rate (kcal/s), number of sucks per burst (n), inter-burst intervals (s), and inter-suck intervals (s). On this platform, a separate entry for the eleven microstructural parameters is not done to avoid redundancy in the description. The study focuses on comparing these parameters between males and females to understand the influence of biological sex on ingestive behavior.
Cluster identification | Five years after bariatric surgery
  Identification of clusters of good and poor response to RYGB five years after surgery based on the variance of the single microstructural parameters of ingestive behaviour
Correlation of Percentage Excess Body Mass Index Loss with the Microstructural Parameters of Ingestive Behaviour Measured with the Drinkometer Device Five Years After Roux-en-Y Gastric Bypass Surgery | Five years after bariatric surgery
  This study aims to investigate the correlation between percentage excess body mass index (BMI) loss (%EBMIL) and microstructural parameters of ingestive behavior, measured using the Drinkometer device, five years after Roux-en-Y gastric bypass (RYGB) surgery. The eleven microstructural parameters considered are: mean suck energy intake (kcal), mean suck duration (s), mean suck rate (kcal/s), mean suck maximal rate (kcal/s), burst number (n), burst energy intake (kcal), burst duration (s), burst rate (kcal/s), number of sucks per burst (n), inter-burst intervals (s), and inter-suck intervals (s).
  This study explores how these microstructural parameters of ingestive behavior correlate with the long-term success of RYGB surgery as indicated by %EBMIL. By understanding these correlations, we aim to gain insights into the behavioral mechanisms that contribute to the maintenance of weight loss post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Bueter, MD, DPhil, Principal Investigator — University of Zurich
Locations (2):
- Switzerland (2):
  - Hospital Männedorf, Männedorf, Canton of Zurich
  - University Hospital Zurich, Department of Surgery and Transplantation, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gero D, Steinert RE, le Roux CW, Bueter M. Do Food Preferences Change After Bariatric Surgery? Curr Atheroscler Rep. 2017 Sep;19(9):38. doi: 10.1007/s11883-017-0674-x. PMID 28779431
- [Background] le Roux CW, Bueter M. The physiology of altered eating behaviour after Roux-en-Y gastric bypass. Exp Physiol. 2014 Sep;99(9):1128-32. doi: 10.1113/expphysiol.2014.078378. PMID 25210112
- [Background] Gero D, File B, Alceste D, Frick LD, Serra M, Ismaeil AE, Steinert RE, Spector AC, Bueter M. Microstructural changes in human ingestive behavior after Roux-en-Y gastric bypass during liquid meals. JCI Insight. 2021 Aug 9;6(15):e136842. doi: 10.1172/jci.insight.136842. PMID 34369388
- [Background] Alceste D, Serra M, Raguz I, Gero D, Thalheimer A, Widmer J, File B, Ismaeil A, Steinert RE, Spector AC, Bueter M. Association between microstructure of ingestive behavior and body weight loss in patients one year after Roux-en-Y gastric bypass. Physiol Behav. 2022 May 1;248:113728. doi: 10.1016/j.physbeh.2022.113728. Epub 2022 Feb 5. PMID 35134394
- [Background] Lutz TA, Bueter M. Physiological mechanisms behind Roux-en-Y gastric bypass surgery. Dig Surg. 2014;31(1):13-24. doi: 10.1159/000354319. Epub 2014 May 8. PMID 24819493
- [Background] Gero D, File B, Justiz J, Steinert RE, Frick L, Spector AC, Bueter M. Drinking microstructure in humans: A proof of concept study of a novel drinkometer in healthy adults. Appetite. 2019 Feb 1;133:47-60. doi: 10.1016/j.appet.2018.08.012. Epub 2018 Sep 1. PMID 30179650
- [Background] Serra M, File B, Alceste D, Raguz I, Gero D, Thalheimer A, Widmer J, Ismaeil A, Steinert RE, Spector AC, Bueter M. Burst-pause criterion derivation for drinkometer measurements of ingestive behavior. MethodsX. 2022 May 11;9:101726. doi: 10.1016/j.mex.2022.101726. eCollection 2022. PMID 35620756